CLINICAL TRIAL: NCT02356861
Title: LED Light Therapy to Improve Cognitive/Psychosocial Function in TBI-PTSD Veterans
Brief Title: LED Light Therapy to Improve Cognitive & Psychosocial Function in TBI-PTSD Veterans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: manufacturer of the 1-of-a-kind, proprietary Treatment device went out of business. Tx. could not be delivered (see final report)
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D1768-P; 1I21RX001768-01 (NIH)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury (TBI); Post-traumatic Stress Disorder (PTSD)
Keywords: treatment; photobiomodulation; Veterans; brain-injury; TBI; PTSD
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the design included double blind procedures for study staff and participants. study devices were be: 1) an active LED helmet that delivered therapeutic frequencies of light and 2) and identical helmet in all ways except it did not deliver therapeutic frequencies of light
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real, Active LED Treatment Series (Active Comparator): These participants will first receive a series of 12, sham LED treatments, At 1 week post completion of the Sham LED treatment series, participants in this group receive a series of 12 real LED treatments from the helmet housing LEDs that deliver photons of light in the infrared range.
  Interventions: Device: Photomedex Sham Helmet with Red/Near-Infrared Light-Emitting Diodes (LEDs) that are not turned on
- Sham LED Treatment Series (Sham Comparator): These participants will first receive an initial series of 12 sham LED treatments from the helmet containing the sham LEDs.
  Interventions: Device: Photomedex Sham Helmet with Red/Near-Infrared Light-Emitting Diodes (LEDs) that are not turned on

INTERVENTIONS:
Device: Photomedex Sham Helmet with Red/Near-Infrared Light-Emitting Diodes (LEDs) that are not turned on — The LED helmet from Photomedex, Montgomeryville, PA will be used.
  18 LED pods are in the helmet. Each LED pod:
  Pod size: 19 cm2 Power output: 692.5 mW Power density: 36.5 mW/cm2
  20 NIR diodes, 830 nm and 4 red diodes, 633 nm.
  1 J/cm2 = 30.4 sec

SUMMARY:
The purpose of this study is to learn if an experimental treatment can help thinking ability, and memory in Veterans with mild or moderate traumatic brain injury (mTBI), and post-traumatic stress disorder (PTSD). The experimental treatment is called transcranial, light-emitting diode (LEDs) therapy,and uses groups of LEDs mounted inside a helmet. The helmet is worn on the head, and the LEDs shine painless light on the sides, middle and front of the head through the scalp. The participants receive a series of LED treatments which take place as outpatient visits at the VA Boston Healthcare System, Jamaica Plain Campus. The LEDs contain near-infrared diodes. The FDA considers the LED device used here, to be a non-significant risk device. The LEDs do not produce heat.

DETAILED DESCRIPTION:
Rationale:

The rational for using near-infrared LEDs is two-fold: 1) These wavelengths have been shown to improve adenosine triphosphate (ATP) production, especially in hypoxic or compromised cells. 2) Recent studies in humans have also shown an increase in regional cerebral blood flow subjacent to where the near-infrared LEDs were placed on the scalp (Schiffer et al., 2009; Nawashiro et al., 2012).

General Explanation of the Light-Emitting Diode (LED) Treatment Procedure:

The LED treatments take place as outpatient visits at the VA Boston Healthcare System (VABHS) Jamaica Plain Campus (JP Campus), 150 South Huntington Ave., Boston, MA, 02130.

The Transcranial LED treatment procedure is painless, non-invasive and no heat is generated. It involves placing a lightweight helmet on the head. The helmet contains some light-emitting diodes (LEDs). The LEDs are not visible (near-infrared wavelengths of light).

During some of the LED treatments, the lights are turned on. During some of the LED treatments, the lights are not turned on. All participants who are part of this study will receive some LED treatments when the LED lights are turned on.

The participant will not feel anything when the LED lights are on; it is a painless, noninvasive treatment procedure. There are small fans built into the LED helmet (to assist in circulating air inside the helmet and help with cooling). The participant will always hear the fans, during each LED treatment, whether the LEDs are on, or they are not on.

There are 3 sequential parts to each LED treatment visit, while the LED helmet is on the head:

Part 1: The LEDs in the center of the helmet are on for 6 and a half minutes; then turned off.

Part 2: The LEDs in the right side of the helmet are on for 6 and a half minutes; then off.

Part 3: The LEDs in the left side of the helmet are on for 6 and a half minutes; then off.

The entire treatment with the LED helmet in place on the head is about 20 minutes, per treatment visit. There is no potential for eye damage, because LED light is not a laser light.

The participant will remain in street clothes, and will be treated in a soft recliner chair. Each visit lasts about 35 to 45 minutes, allowing time for record keeping.

No liquids or gel are used to hold the LEDs in place on the head. Each participant will be provided with his/her own clear plastic liner for the LED helmet. This clear plastic liner will be assigned to each participant, and only used by that participant. It will be kept in a locked filing cabinet in the treatment room, and discarded after the participant's completion of the study.

There are 12 visits in each LED treatment series; and each participant will participate in two LED treatment series. Each LED treatment series lasts for 6 weeks. Each LED treatment visit is scheduled twice per week, with at least 48 hours between each visit.

All appointments are scheduled ahead, for a specific day and time of day, at the convenience of the participant. If the participant needs to miss an appointment, that appointment will be re-scheduled. However, if the participant misses more than 1 appointment in a row, over a two-week period, he/she will be withdrawn from the study. This is because it is very important to treat at least two times per week for the 6 weeks, until all 12 LED treatments have been completed, in each of the two LED treatment series.

The length of time for participation in the actual treatment portion of this study is 3 months (two treatment periods of about 1.5 months, each). The total time of participation including pre- testing, and final follow-up testing at 2 months after the last LED treatment visit, is about 5 months.

This study is sponsored by the Department of Veterans Affairs, Clinical Science Research and Development. There are no potential conflicts of interest associated with this research.

Referral and Screening of Potential Participants:

After self-referral to this study, each potential participant is contacted by telephone, and a description of the full study protocol is explained, including the time required, and reimbursement for time and effort. After the initial contact by telephone, an initial visit to the VABHS, JP campus may be scheduled with Dr. Knight, the PI, or someone on his staff. At this time, the entire study will be explained and questions answered. If the potential participant wishes to do so, he/she may sign the Informed Consent Form (ICF) at this first visit.

After the ICF has been signed, an appointment is then scheduled for Neuropsychological Screening testing. These tests measure the ability to think and remember recent information. If results from the Neuropsychological Screening tests show that the potential participant is eligible for entry into this study, an additional appointment is scheduled where Additional Neuropsychological Testing is performed, and Additional Health Information is obtained.

The Additional Neuropsychological Tests also measure the ability to think and remember recent information. These tests take place at the VABHS, JP. They are administered by Dr. Knight or his staff, and they require a two-hour visit.

During the same two-hour visit, Additional Health Information (paper and pencil) is acquired in the following areas: 1) any pain experienced on a regular basis; 2) fatigue that is experienced on a regular basis; and 3) questions regarding health - for example, how often in the past 30 days symptoms may have been present from each of nine body systems: cardiac, pulmonary, dermatological, gastrointestinal, genitourinary, musculoskeletal, neurological, and psychological.

The Additional Neuropsychological Tests (and the Additional Health Information) are each acquired four times during participation in the study:

Time 1) Within 1 or 2 weeks before the 1st LED Treatment

Time 2) Within 1 week after the 12th LED treatment in the First Series of LED Treatments

Time 3) Within 1 week after the 12th LED treatment in the Second Series of LED Treatments

Time 4) At 2 months after the 12th LED treatment in the Second Series of LED Treatments

In summary, there are a total of 4 visits for the areas of "Additional Neuropsychological Tests and Additional Health Information,"

Statistical Analyses and Power Statement:

There will be one group of 50 participants recruited. Each will serve as his/her own control in this within-subject, repeated measurement partial crossover design.

A score for each of 3 cognitive domains will be analyzed pre- and post- LED intervention:

1. Attention/Executive Function: Digit Span Subtests (WAIS-IV; Wechsler, 2008); Trail-Making Test (Delis, Kaplan, Kramer, 2001); and Stroop Test ("Color-Word" test) (Delis, Kaplan, Kramer, 2001)
2. Learning and Memory: California Verbal Learning Test-II (CVLT-II; Delis, Kramer, Kaplan, & Ober, 2000)
3. Psychomotor/Visual Spatial; Continuous Performance Test (Administered on computer; RVisual CPT, NES3) (Letz & Baker, 1988; Rosvold et al., 1956); Rey Osterrieth Complex Figure Test (ROCF) (Knight & Kaplan, 2004)

Power Analysis:

Power was computed under the following assumptions for ANOVA: a) alpha = .05 (1-tail); b) to establish clinical relevance, Cohen's large effect size (.25) was used. Power = .86 to detect a significant between-group difference in change from Baseline to end of Treatment for an interim analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

The participants for this study will be recruited from flyers posted within the VA Boston Healthcare System and Veterans who contact the study after hearing about it from an outside referral source who knows that the study is actively recruiting participants. Participants must have both mild or moderate TBI and PTSD

* Males or Females; Ages 18 - 65 years old
* Must live within 50 miles of and be physically able to travel to the VA Boston Healthcare System, Jamaica Plain, for Neuropsychological testing and transcranial LED treatments
* Must meet screening criteria from the Neuropsychological Screening Tests
* Must meet screening criteria for a PTSD diagnosis

Exclusion Criteria:

Exclusion Criteria:

* Not meeting criteria for post-traumatic stress disorder and for mild or moderate traumatic brain injury
* Had Gulf War Veterans' Illnesses (GWVI), but did not answer 'Yes' to the following questions: 1) Difficulty concentrating and/or 2) Difficulty remembering recent information, on the Symptom Questionnaire
* Less than age 18, or greater than age 60
* Presence of a neurodegenerative disease such as Amyotrophic Lateral Sclerosis (ALS), Parkinson's, Dementia
* Presence of a life-threatening disease such as cancer
* Presence of a severe mental disorder such as schizophrenia, or severe depression
* Physical limitations that would prevent traveling to the VA Boston Healthcare System, Jamaica Plain, for Neuropsychological testing and transcranial LED treatments
* Current substance abuse or in active treatment
* Did not meet screening criteria from the Neuropsychological Screening Tests
* does not reside physically within 50 miles of the VA Boston - Jamaica Plain VA Hospital location

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Stroop Test ("Color-Word" test) (Delis, Kaplan & Kramer, 2001) | 1 Week after the last LED treatment in each treatment series
  Attention/Executive Function

SECONDARY OUTCOMES:
Digit Span Subtests (WAIS-IV; Wechsler, 2008) D-KEF Trails (Delis, Kaplan & Kramer, 2001) | 1 Week after the last LED treatment in each treatment series
  Additional Attention/Executive Function
California Verbal Learning Test-II (CVLT-II; Delis, Kramer, Kaplan, & Ober, 2000) | 1 Week after the last LED treatment in each treatment series
  Learning and Memory
Beck Depression inventory (BDI; Beck, 2006) | 2 Months after the last LED treatment
  Mood [ Time Frame:
hort Form-36V Plus (Ware et al., 2000) Health Symptom Checklist (HSC). | 2 Months after the last LED treatment
  Data for General Physical Health. The HSC is a comprehensive list of 34 frequently reported health and mental health symptoms originally adapted from Bartone et al., (1989). It asks how often in the past 30 days each of the health symptoms was experienced. Symptoms from nine body systems are assessed (cardiac, pulmonary, dermatological, gastrointestinal, genitourinary, musculoskeletal, neurological, and psychological).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Knight, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No